CLINICAL TRIAL: NCT07184294
Title: Assessing the Feasibility of Different Types of Massage to Reduce Anxiety During Chemotherapy Infusion
Brief Title: Different Types of Massage Therapy to Reduce Anxiety During Chemotherapy Infusion in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24302; NCI-2025-06187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24302 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (FL, HNS, HA, combination, no massage) (Experimental): Patients receive massage therapy according to a randomized schedule to the FL, HNS, hands/arms (HA), combination of all three groups (FL, HNS, HA) or no massage therapy over 30 minutes over 5 chemotherapy sessions total on study. Patients also undergo saliva sample collection on study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Massage Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive no massage therapy
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo saliva sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Massage Therapy — Receive FL therapy
  Other Names: Massage
Procedure: Massage Therapy — Receive HNS therapy
  Other Names: Massage
Procedure: Massage Therapy — Receive HA therapy
  Other Names: Massage
Procedure: Massage Therapy — Receive combination FL, HNS, and HA therapy
  Other Names: Massage
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well different types of massage therapy works to reduce anxiety during chemotherapy infusions in patients with cancer. Many cancer patients experience moderate to severe anxiety and anxiety can worsen by the anticipation of medical procedures that patients have to receive, particularly chemotherapy. Massage therapy, as a complementary treatment, has shown promise in lessening both physical and psychological symptoms associated with cancer and its treatments. Research has also shown the benefits of massage therapy in reducing pain, stress, anxiety, nausea (upset stomach), fatigue (tiredness), and depression in cancer patients. Different types of massage therapy may potentially reduce some cancer patients' symptoms, enhance their treatment, and reduce treatment related side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of 30-minute massages targeting various body regions among patients with cancer receiving anticancer therapy infusion.

II. Assess which type of massage is preferred by patients with cancer receiving anticancer therapy infusion.

SECONDARY OBJECTIVE:

I. To assess the change in anxiety levels after each type of massage therapy during infusion.

EXPLORATORY OBJECTIVE:

I. To evaluate changes in other symptoms, such as: pain, fatigue, nausea, depression, and overall well-being, using data obtained from the Edmonton Symptoms Assessment scale (ESAS) after each type of massage therapy.

OUTLINE:

Patients receive massage therapy according to a randomized schedule to the feet/legs (FL), head/neck/shoulder (HNS), hands/arms (HA), combination of all three groups (FL, HNS, HA) or no massage therapy over 30 minutes for 5 chemotherapy sessions total on study. Patients also undergo saliva sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older at time of consent
* The study is open to all participants regardless of gender, race, or ethnicity
* Participants should have had at least 1 cycle of the chemotherapy regimen at the time of recruitment
* Participant must have a baseline anxiety score > 3 on the Visual Analog scale (VAS)
* Scheduled for at least six more infusion sessions
* Participant has had complete blood count (CBC) lab work completed in the past 24 hours

Exclusion Criteria:

* Platelet count less than 20,000. Patients taking anticoagulants are not excluded, as the protocol for massage in infusion ensures that deep pressure massage is never performed, and patient's massage will not exceed a 3 on the Walton scale
* Absolute neutrophil count (ANC) less than 500
* Patient has received radiation therapy to any of the targeted areas within the past 90 days
* Any patient that is currently using a cold therapy device that would interfere with their ability to have a massage without removing the device (cold gloves, cold socks)
* Had surgery on their foot, leg, head, neck, shoulder, hands, or arms within the past three months
* Participant has rashes, open wounds, or any skin conditions that could be exacerbated by massage
* Known allergies to creams, lotions, or any other substances that may be used during the massage therapy sessions
* Ongoing uncontrolled active psychiatric condition that would interfere in the conduct of the study (e.g., mood disorders, anxiety, psychosis disorders, or substance use), as determined by the patient's primary cancer team
* Participants with a known allergy to Bioton dual-purpose massage cream or any of its ingredients will be excluded from the study
* In order to minimize undue influence and coercion, the study team will not personally solicit an employee for participation: An employee who is under the direct/indirect supervision of the principal investigator (PI)/a co-investigator/the study manager and a direct study team member
* Pregnancy
* Any participants with bone metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Participation rate | Up to 1 year
  Will consider the study feasible if >=70% of patients are able to complete the massage intervention at each session. Descriptive summary will be provided (including 95% confidence intervals [CI]).
Completion rate | Up to 1 year
  Descriptive summary will be provided (including 95% CI).

SECONDARY OUTCOMES:
Change in anxiety levels (State-Trait Anxiety Inventory) | Up to 1 year
  Will be assessed by the items from the State-Trait Anxiety Inventory. Will use paired t-tests to assess the impact of each massage intervention, by comparing changes in outcome measures from pre to post intervention within each session. Second, will apply mixed effect models to evaluate the main effects of interventions and time points (and their interaction) on the changes in outcome measures, while accounting for the individual differences, session variability, as well as missing data. These analyses will provide estimates and effect sizes to help inform the design of future studies. They are intended to detect a signal rather than test a formal hypothesis.
Change in anxiety levels (Edmonton Symptom Assessment System) | Up to 1 year
  Will be assessed by the items from the Edmonton Symptom Assessment System. Will use paired t-tests to assess the impact of each massage intervention, by comparing changes in outcome measures from pre to post intervention within each session. Second, will apply mixed effect models to evaluate the main effects of interventions and time points (and their interaction) on the changes in outcome measures, while accounting for the individual differences, session variability, as well as missing data. These analyses will provide estimates and effect sizes to help inform the design of future studies. They are intended to detect a signal rather than test a formal hypothesis.
Change in anxiety levels salivary amylase) | Up to 1 year
  Will be assessed by the items from the salivary amylase. Will use paired t-tests to assess the impact of each massage intervention, by comparing changes in outcome measures from pre to post intervention within each session. Second, will apply mixed effect models to evaluate the main effects of interventions and time points (and their interaction) on the changes in outcome measures, while accounting for the individual differences, session variability, as well as missing data. These analyses will provide estimates and effect sizes to help inform the design of future studies. They are intended to detect a signal rather than test a formal hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope at Irvine Lennar, Irvine, California, United States